CLINICAL TRIAL: NCT04200248
Title: A Multi-Center, Randomized, Double Masked and Active Controlled Phase II Study Assessing the Efficacy and Safety of Intravitreal Injections of RBM-007 Monotherapy and RBM-007 in Combination With Eylea® Compared to Eylea® Monotherapy
Brief Title: A Phase II Study of RBM-007 Alone and RBM-007 With Eylea® in Subjects With Wet Age-related Macular Degeneration
Acronym: TOFU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ribomic USA Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RBM 007-002
Record Dates: First submitted 2019-12-08; First posted 2019-12-16 (Actual); Results first posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-04

CONDITIONS: Exudative Age-related Macular Degeneration
Keywords: Fibrosis; Edema; Neovascularization
MeSH Terms: conditions — Fibrosis; Edema; Neovascularization, Pathologic | interventions — aflibercept; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sham + RBM-007 (Experimental): Sham + RBM-007 intravitreal injection
  Interventions: Drug: RBM-007 Injectable Solution; Drug: Sham
- RBM-007 + Aflibercept (Experimental): RBM-007 + Aflibercept intravitreal injection
  Interventions: Drug: RBM-007 Injectable Solution; Drug: Aflibercept
- Sham + Aflibercept (Active Comparator): Sham + Aflibercept intravitreal injection
  Interventions: Drug: Aflibercept; Drug: Sham

INTERVENTIONS:
Drug: RBM-007 Injectable Solution — RBM-007 Injectable Solution
  Arms: RBM-007 + Aflibercept; Sham + RBM-007
Drug: Aflibercept — EYLEA® (aflibercept) Injection, for Intravitreal Use
  Arms: RBM-007 + Aflibercept; Sham + Aflibercept
Drug: Sham — Sham intravitreal injection
  Arms: Sham + Aflibercept; Sham + RBM-007

SUMMARY:
This is a multicenter, active-controlled, double masked study assessing the safety, efficacy and durability of four monthly intravitreal (IVT) injections of RBM-007 monotherapy, and four monthly RBM-007 injections in combination with Eylea® dosed at every other month, compared to Eylea® monotherapy dosed at every other month in approximately eighty-one subjects with exudative age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
RBM-007 is a novel oligonucleotide-based aptamer having potent anti-FGF2 activity and anti-VEGF-expression activity

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed written informed consent.
2. Male or female 55 years of age or older on the date of signing the consent and able and willing to comply with all treatment and study procedures.
3. Diagnosis of exudative age-related macular degeneration in the study eye, for which previous standard treatment with intravitreal anti-vascular endothelial growth factor agents (at least 4 injections over the past 8 months) has demonstrated incomplete resolution of exudation, as assessed by spectral domain optical coherence tomography.
4. Presence of macular edema or subretinal fluid.
5. Absence of central atrophy or retinal epithelial tear in the fovea or any condition preventing visual acuity improvement in the study eye.
6. Visual acuity of 78 to 24 letters (20/32 to 20/320) in the study eye.
7. Visual acuity of 24 letters (20/320) or better in the fellow eye.
8. Reasonably clear media and some fixation in the study eye to allow for good quality tomography and fundus photography

Exclusion Criteria:

* Ocular:

  1. Use of any of the following treatments or anticipated use of any of the following treatments to the study eye:

     1. Any intravitreal treatment within 4 weeks prior to Baseline (Visit 1).
     2. Intravitreal or periocular corticosteroid, within 90 days prior to Visit 1 (Day 1) and throughout the study.
     3. Fluocinolone acetonide intravitreal implant, within 12 months prior to Visit 1 (Day 1) and throughout the study.
     4. Visudyne® photodynamic therapy, within 90 days prior to Visit 1 (Day 1) and throughout the study.
  2. Uncontrolled or advanced glaucoma, evidenced by an intraocular pressure of > 21 mmHg or cup/disc ratio > 0.8 while on medical therapy, or chronic hypotony (< 6 mmHg) in the study eye.
  3. Evidence of any other ocular disease other than wet age-related macular degeneration in the study eye that may confound the outcome of the study
  4. History of vitrectomy in the study eye.
  5. Need for ocular surgery in the study eye during the course of the study.
  6. YAG laser capsulotomy within 30 days prior to Visit 1 (Day 1) in the study eye.
  7. Intraocular surgery, including lens removal or laser, within 90 days prior to Visit 1 (Day 1) in the study eye.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Padma Bezwada, Ph.D., Study Director — RIBOMIC USA
Locations (8):
- United States (8):
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Retinal Consultants Medical Group, Sacramento, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Advanced Research, LLC, Coral Springs, Florida
  - Georgia Retina, P.C., Marietta, Georgia
  - Raj K. Maturi, M.D., P.C., Indianapolis, Indiana
  - Valley Retina Institute, PA, McAllen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sham + RBM-007 | RBM-007 + Aflibercept | Sham + Aflibercept
Started | 32 | 31 | 31
Completed | 29 | 28 | 28
Not Completed | 3 | 3 | 3
Not completed — Personal reasons | 0 | 0 | 1
Not completed — Discontinued prior to treatment | 3 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Intent to treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham + RBM-007 | RBM-007 + Aflibercept | Sham + Aflibercept | Total
Number analyzed (Participants) | 32 | 31 | 31 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 0 | 4
  >=65 years | 31 | 28 | 31 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.41 (7.47) | 75.32 (8.64) | 78.52 (7.07) | 78.1 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 15 | 18 | 54
  Male | 11 | 16 | 13 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 6
  Not Hispanic or Latino | 30 | 29 | 29 | 88
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0
  White | 30 | 31 | 31 | 92
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 31 | 31 | 94
Best corrected visual acuity [Mean (Standard Deviation); unit: Letter seen] — Population: Data presented for population treated (8 subjects discontinued before treatment)
  Letter seen
    number analyzed (Participants) | 29 | 28 | 29 | 86
    (all) | 60.24 (13.00) | 66.71 (10.81) | 61.52 (13.83) | 62.78 (13.13)
Central subfield thickness (macula) [Mean (Standard Deviation); unit: Microns] — Population: Data presented for population treated (8 subjects discontinued before treatment)
  Microns
    number analyzed (Participants) | 29 | 28 | 29 | 86
    (all) | 452.07 (138.24) | 398.04 (124.01) | 437.55 (129.34) | 429.58 (131.20)
Macular volume [Mean (Standard Deviation); unit: mm^3] — Population: Measure Analysis Population Description: Data presented for population treated (8 subjects discontinued before treatment)
  mm^3
    number analyzed (Participants) | 29 | 28 | 29 | 86
    (all) | 9.03 (0.23) | 8.84 (0.23) | 9.00 (0.23) | 8.96 (0.23)
Fibrosis [Count of Participants; unit: Participants] — Number of subjects with fibrosis at baseline Population: Measure Analysis Population Description: Data presented for population treated (8 subjects discontinued before treatment)
  Participants
    number analyzed (Participants) | 29 | 28 | 29 | 86
    (all) | 27 | 27 | 28 | 82

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity - Continuous
Description: Mean change in Best Corrected Visual Acuity from Baseline to Week 16
Time Frame: Week 16
Population: Data presented for population treated (8 subjects discontinued before treatment)
Measure: Mean (Standard Error); unit: Letters seen
Arm/Group | Sham + RBM-007 | RBM-007 + Aflibercept | Sham + Aflibercept
Number analyzed (Participants) | 29 | 28 | 29
Letters seen | -6.1 (1.70) | -1.6 (1.75) | 2.4 (1.69)

2. Secondary Outcome: Visual Acuity - Categorical
Description: Percentage of patients gaining >= 15 letters as measured by Best Corrected Visual Acuity from Baseline at Week 16
Time Frame: Week 16
Population: Data presented for population treated (8 subjects discontinued before treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Sham + RBM-007 | RBM-007 + Aflibercept | Sham + Aflibercept
Number analyzed (Participants) | 29 | 28 | 29
Participants | 0 | 0 | 2

3. Secondary Outcome: Macular Thickness Change
Description: Change from Baseline in Central Subfield Thickness by spectral domain optical coherence tomography at Week 16
Time Frame: Week 16
Population: Data presented for population treated (8 subjects discontinued before treatment)
Measure: Mean (Standard Error); unit: microns
Arm/Group | Sham + RBM-007 | RBM-007 + Aflibercept | Sham + Aflibercept
Number analyzed (Participants) | 29 | 28 | 29
microns | 36.5 (12.60) | -5.8 (12.89) | -16.1 (12.55)

4. Secondary Outcome: Macular Volume Change
Description: Change from Baseline in macular volume by spectral domain optical coherence tomography at Week 16
Time Frame: Week 16
Population: Data presented for population treated (8 subjects discontinued before treatment)
Measure: Mean (Standard Error); unit: mm^3
Arm/Group | Sham + RBM-007 | RBM-007 + Aflibercept | Sham + Aflibercept
Number analyzed (Participants) | 29 | 28 | 29
mm^3 | 0.748 (0.120) | 0.0095 (0.124) | -0.010 (0.120)

5. Secondary Outcome: Fibrosis Change
Description: Change from Baseline in sub-retinal hyper-reflective material by spectral domain optical coherence tomography at Week 16
Time Frame: Week 16
Population: Data presented for population treated (8 subjects discontinued before treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Sham + RBM-007 | RBM-007 + Aflibercept | Sham + Aflibercept
Number analyzed (Participants) | 29 | 28 | 29
Participants
  Better | 3 | 8 | 9
  Not better | 26 | 20 | 20

6. Secondary Outcome: Safety - Ocular
Description: Ocular examination (biomicroscopy and ophthalmoscopy) at Week 20 - Number of participants with additional corneal abnormalities
Time Frame: Week 20
Population: Data presented for population treated (8 subjects discontinued before treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Sham + RBM-007 | RBM-007 + Aflibercept | Sham + Aflibercept
Number analyzed (Participants) | 28 | 29 | 29
Participants
  Additional corneal abnormalities | 9 | 11 | 10
  No additional corneal abnormalities | 19 | 18 | 19

ADVERSE EVENTS:
Time Frame: 20 Weeks
Arm/Group | Sham + RBM-007 | RBM-007 + Aflibercept | Sham + Aflibercept
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 2/28 | 2/29 | 1/29
Other Adverse Events (participants affected / at risk) | 15/28 | 17/29 | 8/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham + RBM-007 (N=28) | RBM-007 + Aflibercept (N=29) | Sham + Aflibercept (N=29)
Iritis (Eye disorders) | 2 (2) | 1 (1) | 1 (1)
Vitritis (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Neovascular age-related macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Endophthalmitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham + RBM-007 (N=28) | RBM-007 + Aflibercept (N=29) | Sham + Aflibercept (N=29)
Eye disorders (Eye disorders) | 13 (13) | 15 (15) | 8 (8) — Study eye
Conjunctival haemorrhage (Eye disorders) | 5 (5) | 6 (6) | 3 (3) — Study eye
Dry eye (Eye disorders) | 4 (4) | 1 (1) | 1 (1) — Study Eye
Eye irritation (Eye disorders) | 2 (2) | 2 (2) | 1 (1) — Study eye
Eye pain (Eye disorders) | 2 (2) | 0 (0) | 0 (0) — Study eye

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT04200248/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT04200248/SAP_001.pdf